CLINICAL TRIAL: NCT00695487
Title: Does Intravenous Cannabis Reduce Postoperative Nausea and Vomiting (PONV)?
Acronym: THC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In the intermediate analysis, no effect could be shown, not even a tendency.
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KEK240_07; THC-001
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Nausea; Vomiting
Keywords: Anesthesia; THC; Postoperative Nausea
MeSH Terms: conditions — Nausea; Vomiting; Postoperative Nausea and Vomiting | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Receives 0.125mg/kg THC before emergence
  Interventions: Drug: THC 9-d-tetra hydro cannabinol
- 2 (Placebo Comparator): Receives NaCl before emergence
  Interventions: Drug: THC 9-d-tetra hydro cannabinol

INTERVENTIONS:
Drug: THC 9-d-tetra hydro cannabinol — 0.125mg/kg iv one time

SUMMARY:
The investigators evaluate if intravenously applied THC (Cannabis) reduces postoperative Nausea and vomiting. THC will be given during anesthesia before emergence. We measure how long and how effective it reduces PONV

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* elective open and laparoscopic surgery >1hour

Exclusion Criteria:

* ambulatory surgery
* pregnancy, breast feeding
* >ASA III
* BMI >35
* antipsychotic, antiemetic, cytostatic therapy
* major cardiovascular, renal, hepatic, central nervous system disease
* current chronic cannabis consumption and hard drug abuse
* schizophrenia
* preoperative nausea and vomiting, vestibular disease
* not speaking german or french
* refusal to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Absence of postoperative Nausea and Vomiting | 0-24h after Operation

SECONDARY OUTCOMES:
Psychological and physiological data after ingestion of THC Analgetics required | 0-24h after operation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD, Study Director — Department of Anesthesia, Bern University Hospital , Switzerland
Locations (1):
- Inselspital, Bern University Hospital, Bern, Canton of Bern, Switzerland